CLINICAL TRIAL: NCT05544721
Title: Pre-Operative and Post-Operative Paravertebral Block on Patients With Thoracic Outlet Syndrome.
Brief Title: A Study of Paravertebral Block in Thoracic Outlet Syndrome
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Houssam Farres, M.D., Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 22-006685
Record Dates: First submitted 2022-09-14; First posted 2022-09-16 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Thoracic Outlet Syndrome
Keywords: First rib resection procedure
MeSH Terms: conditions — Thoracic Outlet Syndrome | interventions — Ropivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Paravertebral block pre procedure (Active Comparator): Subjects will receive a preoperative paravertebral block only
  Interventions: Drug: Ropivacaine
- Paravertebral block pre and post procedure (Active Comparator): Subjects will receive one paravertebral block, administered preoperatively and one paravertebral block, administered on postoperative day 1
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Ropivacaine — 0.5% 3-4 mL per level, with levels T1 and T2 will be used as the block injectate

SUMMARY:
This research is being done to evaluate the effects of receiving only a paravertebral block prior to first rib resection procedure versus receiving the block both pre and post procedure.

ELIGIBILITY:
Inclusion Criteria:

- All Thoracic Outlet Syndrome patients scheduled for first rib resection surgery.

Exclusion Criteria:

* Patients who are pregnant.
* Patients with prior first rib resection on side of presentation.
* Patients with complex regional pain syndrome (CRPS).
* Patients with brachial plexus disorder.
* Patients with cervical rib.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-10-05 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Change in pain level | Time of discharge (approximately 1 day), day 1 post-op, day 3 post-op, day 7 post-op, and day 14 post-op
  Measured using the pain visual analog scale (VAS). The VAS line will be 100 mm long with each end marked with "no pain" on the left, and "worst possible pain" on the right; participant identify their pain level by indicating a point on the line between each end and this point is measured from the "No pain" end, and the number of millimeters is reported as the pain score.

SECONDARY OUTCOMES:
Change in quality of life | Time of discharge (approximately 1 day), day 1 post-op, day 3 post-op, day 7 post-op, and day 14 post-op
  Measured using the Short Form (SF-36) Health Survey; The SF-36 Health Survey is a 36-item, participant-reported survey that measures patient health and disability. Possible scores range from 0 to 100, with 0 indicating maximum disability, and 100 indicating no disability
Length of stay | Approximately 1 day
  Number of hours subjects are in the hospital following their surgical procedure

CONTACTS AND LOCATIONS:
Overall Officials: Houssam Farres, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials